CLINICAL TRIAL: NCT05652231
Title: Assessment of Dental Caries Among a Group of Institutionalized Orphan Children Compared to Parented School Children
Status: Completed | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mennat Allah Ashraf A.Elsabour, Primary Investigator, Ahram Canadian University
Other Study IDs: ACU 111
Record Dates: First submitted 2022-12-06; First posted 2022-12-15 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- School children (control group): parented school children (control group)
  Interventions: Diagnostic Test: caries assessment
- Non-Governmental orphanage children (exposed group 1)
  Interventions: Diagnostic Test: caries assessment
- Governmental orphanage children (exposed group 2)
  Interventions: Diagnostic Test: caries assessment

INTERVENTIONS:
Diagnostic Test: caries assessment — the child will examined for dental caries, caries prevalence, caries indices (def and DMF, or DMF)

SUMMARY:
Children from two orphanages will be examined for dental caries experience, in comparison to parented school children.

DETAILED DESCRIPTION:
A total of 156 children were included in this study, they were, residing in governmental orphanage, non-governmental orphanage and parented children attending primary school. Written informed consent was obtained prior to the start of the study, form legal guardians or child's parent. Dental examination was carried out on an ordinary chair beside a window on day light. DMF and def indices were used to assess dental caries for primary and permanent teeth. Also, unmet treatment need index, care index and significant caries index were calculated.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy children aged from six to12 years old

Exclusion Criteria:

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: apparently healthy children aged from six to12 years old
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
caries experience | baseline record
  measured using DMF/ def index

CONTACTS AND LOCATIONS:
Locations (1):
- Ahram Canadian University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khattab NMA, Abd-Elsabour MAA. Assessment of dental caries among a group of institutionalized orphan children compared to parented school children: case-control study. BMC Oral Health. 2023 Apr 5;23(1):202. doi: 10.1186/s12903-023-02915-1. PMID 37020200